CLINICAL TRIAL: NCT01813747
Title: Mandible and Sub-mandible Using the 1440nm Wavelength Laser and Hand Piece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN10-DS-MS2
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Skin Tightening of the Mandibular and Sub-mandibular Areas

STUDY DESIGN:
Intervention Model Description: Even though this study has recruited slightly more than 10 participants, it is a feasibility study, designed to test the prototype rather than measuring health outcomes. It is to confirm the operating specifications before beginning a full clinical trial.
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1440 nm wavelength laser with hand piece (Experimental): To assess the effectiveness of the 1440 nm wavelength laser with handpiece for skin tightening and laser lipolysis for the mandibular and sub-mandibular areas
  Interventions: Device: 1440 nm wavelength laser with handpiece (Cynosure)

INTERVENTIONS:
Device: 1440 nm wavelength laser with handpiece (Cynosure) — To assess the effectiveness of device in skin tightening and laser lipolysis in the mandibular and sub-mandibular areas.

SUMMARY:
The purpose of this study is to use the 1440nm Wavelength laser along with the hand piece to provide clinical outcome data for treatment of the mandibular and submandibular areas specifically for skin tightening and laser lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects 18-65 years of age
* Presents for treatment of their unwanted skin laxity and fat in the mandibular and submandibular areas for an improved aesthetic appearance and is willing to undergo laser treatment
* Understands/accepts obligation not to receive any other procedures in the mid-face to sub-mandibular areas through 3 months follow up visit
* Understands/accepts the obligation and is logistically able to present for all scheduled follow up visits
* Is capable of understanding the consent form and able to provide written consent to participate in the study and any other practice consents for anesthesia and surgical procedures
* Understands/accepts obligation to have facial photographs taken
* Understands/accepts may be asked to consent to having a two 2mm biopsies in an inconspicuous place such as behind the ear
* Agrees to maintain present diet and exercise program

Exclusion Criteria:

* Has had any procedure in the mid-face to sub-mandibular areas in the last six months
* Has a history of thrombophlebitis, history of coagulation disorders or using anticoagulant medications
* Has a significant systemic illness or immunity disorder or localized condition affecting treatment area
* Is female and pregnant, was pregnant or given birth within the last three months, is currently breast feeding, or planning a pregnancy during the course of the study
* Has known history of allergic reactions to local anesthesia
* Has any other medical condition, that, in the investigator's opinion would interfere with the subject's participation in the study
* Is susceptible to light induced seizures or history of seizures
* Has a history of keloid formation
* Has therapies or medications which may interfere with the treatment (including medications causing photosensitivity
* Has a BMI above 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluation | 3 months post last treatment
  Photos will be evaluated by the investigator comparing time baseline and 3 month photos using the global aesthetic improvement scale
Photographic Evaluation | 3 months post last treatment
  Photographs will be evaluated and compared by investigator for baseline and 3 month images using the Cervicomental Angle Scale

SECONDARY OUTCOMES:
Number of participants with adverse events | up to 3 months post last treatment
  Side effects and events will be recorded
Photographic Evaluation | 1 week post treatment
  Photos will be evaluated by the investigator comparing time baseline and 1 week photos using the global aesthetic improvement scale
Photographic Evaluation | 1 week post treatment
  Photographs will be evaluated and compared by investigator for baseline and 1 week images using the Cervicomental Angle Scale

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Cosmetique - Dermatology, Laser & Plastic Surgery LLP, Greenvale, New York, United States